CLINICAL TRIAL: NCT02133651
Title: Characterization of the Microbial Genomics of Fecal Bacteriotherapy (FBT): Intestinal Microbiota Transplantation (IMT) for Recurring Clostridium Difficile
Brief Title: Mucosal Versus Fecal Microbiota in FMT
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Colleen S Kraft MD, Assistant Professor, Emory University
Other Study IDs: IRB00069524
Record Dates: First submitted 2014-05-05; First posted 2014-05-08 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile; Intestinal Microbiota Transplantation; Diarrhea; Fecal Microbiota Transplant
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal matter from the consented donor, consented recipient at 3 time points will be stored in a -80 freezer.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clostridium difficile infection is the most common cause of antibiotic-associated diarrhea. Treatment of this infection usually occurs using other antibiotics, but many individuals have persistent diarrhea and multiple relapses. Fecal Transplant (FMT), or Intestinal Microbiota Transplantation, (IMT) has been shown to be efficacious when administered after treatment for C. difficile. This study will involve taking biopsies from patients during their FMT/IMT via colonoscopy, and determine if there are differences in the mucosal flora as compared to the stool flora. The investigators hope to discover the critical parts of a healthy microbiota.

DETAILED DESCRIPTION:
A total of 20 subjects with at least one relapse of Clostridium difficile infection undergoing Intestinal Microbiota Transplantation via colonoscopy will be recruited in this study. The patients will produce a stool specimen at the time of colonoscopy and a biopsy will be obtained during the colonoscopy. At 2 weeks and 10 weeks, stool specimens and anoscopy will be collected to be tested for C. difficile polymerase chain reaction (PCR) and the fecal microbiota. Subjects will be referred from all locations of Emory Healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient or outpatient adults, age ≥18
* Have had at least 1 relapse of C. difficile
* Patients who have had previous FMT

Exclusion Criteria:

* Pregnant or breastfeeding
* Critically or acutely ill (Fever will be defined as a documented temperature >37.8°C)
* Ileus or toxic megacolon
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Clostridium difficile infection at least twice and will be undergoing intestinal microbiota transplantation (IMT) via a colonoscopy for treatment from Emory University Hospital and Emory University Midtown.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who experience resolution of diarrhea associated with C. difficile infection without relapse 2 weeks and 10 weeks post Intestinal Microbiota Transplantation (IMT) | 10 weeks post IMT

CONTACTS AND LOCATIONS:
Overall Officials: Colleen S. Kraft, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Friedman-Moraco RJ, Mehta AK, Lyon GM, Kraft CS. Fecal microbiota transplantation for refractory Clostridium difficile colitis in solid organ transplant recipients. Am J Transplant. 2014 Feb;14(2):477-80. doi: 10.1111/ajt.12577. Epub 2014 Jan 16. PMID 24433460